CLINICAL TRIAL: NCT01841138
Title: Changes of Serum Electrolytes During Bowel Prep With PEG 3350 + Ascorbic Acid - a Prospective Study
Status: Completed | Type: Observational
Sponsor: Klinik Bogenhausen (Other)
Responsible Party: Principal Investigator, Arne Schneider, PI, Klinik Bogenhausen
Other Study IDs: GastroKMBColEl
Record Dates: First submitted 2013-01-31; First posted 2013-04-26 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Colonoscopy
Keywords: colonoscopy; bowel preparation; electrolytes; osmolality; water

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: Patients who undergo bowel preparation with PEG 3350 + ascorbic acid may have significant changes of serum electrolytes.

A new PEG solution (Moviprep = PEG 3350 + ascorbic acid) for colonoscopy reduces the amount of cathartic solution to 2 liters, but requires drinking of additional liquid for optimal results. Ingestion of a high volume of free water bears a risk for severe changes of serum electrolytes, particularly for sodium and potassium.

In this trial, patients undergo regular bowel preparation for standard colonoscopy with Moviprep (2 liters Moviprep split-dose plus ≥2 liters of free liquid until sufficient cleansing is achieved). Blood samples for serum sodium, potassium, chloride, magnesium, phosphate, calcium and serum osmolarity are taken before the beginning of the prep procedure and right before colonoscopy. The interval between both blood samples that will be compared is roughly 24 hours. Additionally, the volume of prep solution and additional liquid is recorded. The quality of bowel preparation is visually rated during colonoscopy with a validated score.

Pre- and postpreparation serum parameters will be compared. Primary outcome measure is the proportion of patients who have a serum sodium beyond the reference values after the completion of bowel preparation. Secondary outcome parameters are the proportion of patients with other serum electrolytes or serum osmolarity beyond the reference. Moreover, changes of serum electrolytes and osmolarity will be correlated with the amount of prep solution and liquid.

ELIGIBILITY:
Inclusion Criteria:

* indication for colonoscopy
* >=18 years

Exclusion Criteria:

* <18 years
* acute inflammatory bowel disease
* previous bowel resection
* high-grade cardiac or renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indicaton for colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2010-07; Primary Completion 2015-12 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with serum sodium concentration beyond the limits of normal after the completion of bowel preparation | within 2 hours before the beginning of colonoscopy

SECONDARY OUTCOMES:
Proportion of patients with serum potassium or calcium or chloride or magnesium concentration beyond the limits of normal after the completion of bowel preparation | within 2 hours before the beginning of colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Bogenhausen - Klinikum München GmbH, Munich, Germany